CLINICAL TRIAL: NCT02654340
Title: Biomarkers for Tuberous Sclerosis Complex: An International Multicenter Observational Longitudinal Protocol
Brief Title: Biomarkers for Tuberous Sclerosis Complex (BioTuScCom)
Acronym: TuScCom
Status: Terminated | Type: Observational
Why Stopped: Study no longer pursued.
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: TSC 08-2018
Record Dates: First submitted 2015-10-13; First posted 2016-01-13 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Hypomelanotic Macules; Facial Angiofibroma; Shagreen Patches; Ungual Fibromas; Cortical Dysplasia; Cardiac Rhabdomyoma; Lymphangioleiomyomatosis; Renal Angiomyolipoma; Subependymal Giant Cell Astrocytoma
Keywords: Tuberous sclerosis complex; Biomarker
MeSH Terms: conditions — Tuberous Sclerosis; Malformations of Cortical Development; Lymphangioleiomyomatosis; Angiomyolipoma; Astrocytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample applied on the Dry Blood Spot (DBS) Filtercard (Centocard®)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Tuberous Sclerosis Complex (TSC): Üarticipants diagnosed with Tuberous Sclerosis Complex (TSC) aged between 2 months and 50 years.

SUMMARY:
International, multicenter, observational, longitudinal study to identify biomarker/s for Tuberous Sclerosis Complex and to explore the clinical robustness, specificity, and long´-term variability of these biomarker/s

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC) is an autosomal dominant genetic disorder characterized by the growth of numerous tumors in different body parts related to dysregulation of the mechanistic target of rapamycin (mTOR) pathway. The overall incidence of TSC is estimated to be as high as 1 in 6000 to 10,000 live birth.The main aspects of TSC that influence the quality of life are associated with the brain: seizures, evelopmental delay, intellectual disability, and autism. However, the incidence and severity of the various aspects of TSC can vary widely.

TSC is generally caused by pathogenic variants in the tumor suppressor genes: TSC1 and TSC2. Confirmation of a clinical diagnosis of tuberous sclerosis is performed via TSC1 and TSC2 sequencing.

There is no cure for TSC, therefore symptomatic therapy is the best possible choice, including mTOR inhibitors, vigabatrin and other antiepileptic drugs for the seizures, and neurosurgery in cases of life-threatening neurological symptoms.

The aim of the study is established TSC specific biomarker/s. Such biomarkers aim to facilitate the diagnosis, treatment personalization and monitoring.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent is obtained from the participant or from the parent / legal guardian
* Participant is aged between 2 and 50 years
* Diagnosis of TSC is genetically confirmed by CENTOGENE

EXCLUSION CRITERIA

* Inability to provide informed consent
* Participant is younger than 2 or older than 50 years
* Diagnosis of TSC is not genetically confirmed by CENTOGENE

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with Tuberous Sclerosis Complex (TSC)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Identification of TSC biomarker/s | 36 months
  All samples will be analyzed for the identification of biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

SECONDARY OUTCOMES:
Exploring the clinical robustness, specificity, and longterm variability of TSC biomarker/s | 36 months
  Samples will be analyzed for the candidate biomarker/s via Liquid Chromatography Multiple Reaction-monitoring Mass Spectrometry (LC/MRM-MS) and compared to merged control, in order to establish the disease-specific biomarker/s. The LC/MRM-MS is performed on an ABSciex 6500 triple quadrupole mass spectrometer, coupled with a Waters Acquity UPLC.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof.Dr, Study Chair — Centogene GmbH
Locations (8):
- University Hospital Center Mother Teresa, Tirana, Albania
- Department of Pediatrics, Alexandria University Children's Hospital, Alexandria, Egypt
- Departmnet of Molecular and Medical Genetics, Tbilisi State Medical University, Tbilisi, Georgia
- Department of Pediatric Genetics, Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala, India
- Rare diseases coordinating centre, Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania
- Departmnet of Pediatric Gastroenterology and Hepatology, The Children's Hospital and Institute of Child Health, Lahore, Pakistan
- Emergency Hospital for Children "Louis Turcanu", Timișoara, Romania
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided